CLINICAL TRIAL: NCT04416997
Title: Hematological Indices in Rheumatoid Arthritis and Its Association With Disease Activity and Severity
Brief Title: Rheumatoid Arthritis Hematological Indices
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Yassine Meligy, Princible investigator, Assiut University
Other Study IDs: HRA
Record Dates: First submitted 2020-05-15; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Rheumatoid Arthritis; Serum Albumin Low
Keywords: Rheumatoid arthritis; Red blood cell distribution; Albumin
MeSH Terms: conditions — Arthritis, Rheumatoid; Hypoalbuminemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood and serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatoid arthritis patients: Blood and serum samples
  Interventions: Procedure: Blood and serum samples

INTERVENTIONS:
Procedure: Blood and serum samples — The blood and serum samples will taken from RA patients

SUMMARY:
Rheumatoid arthritis is a chronic systemic inflammatory and autoimmune disease, characterized by disordered immunity, not regulated cytokines and inflammatory infiltration of the synovial joints. It is the most common inflammatory erosive poly arthritis affecting around 0.5-1% of the worldwide population which leads to joint damage and disability

DETAILED DESCRIPTION:
The etiology of Rheumatoid arthritis is complex, it is established that the gene environmental interaction plays critical roles in the pathology of Rheumatoid arthritis, in addition to smoking, lifestyle, and hormones.

The lesion is mainly concentrated in the synovial tissue, cartilage, and bone. Inflammation is the primary cause of joint deformation and limited joint mobility in Rheumatoid arthritis patients. As the disease progresses, the risk of bone damage and cartilage destruction increases, leading to substantial disability.

The activity of the disease in Rheumatoid arthritis patients is assessed by clinical examination, laboratory tests and radio graphic assessment. Laboratory assessment of Rheumatoid arthritis activity is done routinely by measuring acute phase reactants such as an erythrocyte sedimentation rate and C-reactive protein, which are elevated in active Rheumatoid arthritis patients.

Albumin is the major plasma protein and its determination is used for the prognostic assessment of several diseases. It is a routine marker reflecting both nutritional status and systemic inflammation, and the synthesis of albumin can be suppressed by systematic inflammation and malnutrition.

It was reported that the level of albumin was decreased in Rheumatoid arthritis patients. This low concentration of albumin in Rheumatoid arthritis patients may owing to excessive albumin consumption caused by inflammatory substances.

Red blood cell distribution width is a parameter that reflects the heterogeneity of erythrocyte volume, expressed as the coefficient of variation of red blood cell volume. It is mainly used to differentiate types of anemia. However, some studies have shown that an elevated Red blood cell distribution was positively correlated with the level of inflammation.

Red blood cell distribution was increased in patients with Rheumatoid arthritis, which was associated with inflammation, suggesting that Red blood cell distribution may be a potential auxiliary marker for indicating inflammation process in Rheumatoid arthritis conveniently.

In subjects with articular pain, Red blood cell distribution interpretation is a useful tool in clinical practice to distinguish between articular inflammatory and non-inflammatory joint diseases, as with C-reactive protein. Red blood cell distribution seems to be a surrogate marker of the inflammatory process.

ELIGIBILITY:
Inclusion Criteria:

* Adult RA Patients who fulfilled the 2010 European league against rheumatism criteria for the classification of RA

Exclusion Criteria:1. Individuals with concomitant other autoimmune diseases 2. RA patients with anemia, pregnancy, postpartum, diabetes, obesity hypertension.

3. Patients with age less than 18 years 4. Patients with end stage organ failure.

5. Patients with liver diseases.

6. Patients with hematological disorders.

7. Patients with malignancies

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study will include adult RA patients consecutively presented at the Rheumatology, Rehabilitation and Physical Medicine Department, Assiut University Hospitals from both inpatient department and outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-10-29 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of level of Red blood cell distribution width | Through study completion, an average of 1 year
  Red blood cell distribution width will be measured.
Assessment of level of serum Albumin in Rheumatoid arthritis patients | Through study completion, an average of 1 year
  The level of serum Albumin will be measured in Rheumatoid arthritis patients

SECONDARY OUTCOMES:
The relation between Red blood cell distribution width and level of serum albumin in RA patients and association with the disease activity and severity. | Through study completion, an average of 1 year
  Comparing between the Level of Red blood cell distribution width and level of serum albumin in RA patients, then comparing these results with the other routine parameters of these patients.
  Activity index will be done: Disease activity score (DAS28) DAS28 score of higher than 5.1 is indicative of high disease activity, DAS28 score of higher than 3.2 indicate moderate disease activity whereas DAS28 score below 3.2 indicates low disease activity. Patients are considered to be in remission if they have DAS28 score lower than 2.6 Health assessment questionnaire-disability index (HAQ-DI) will be done, It is used as a subjective measure of physical function of RA patients .There are 20 items in 8 categories: dressing, rising, eating, walking, hygiene, reach, grip, and usual activities.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Meligy, Dr, Principal Investigator — FYMeligy
Locations (1):
- Faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
study the relation between RDW and level of serum albumin in RA patients and association with the disease activity and severity.

REFERENCES:
- [Result] Alpizar-Rodriguez D, Finckh A. Environmental factors and hormones in the development of rheumatoid arthritis. Semin Immunopathol. 2017 Jun;39(4):461-468. doi: 10.1007/s00281-017-0624-2. Epub 2017 Apr 27. PMID 28451785
- [Result] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Ann Rheum Dis. 2010 Sep;69(9):1580-8. doi: 10.1136/ard.2010.138461. PMID 20699241
- [Result] Yan F, Li H, Zhong Z, Zhou M, Lin Y, Tang C, Li C. Co-Delivery of Prednisolone and Curcumin in Human Serum Albumin Nanoparticles for Effective Treatment of Rheumatoid Arthritis. Int J Nanomedicine. 2019 Nov 22;14:9113-9125. doi: 10.2147/IJN.S219413. eCollection 2019. PMID 31819422